CLINICAL TRIAL: NCT06860750
Title: A Randomized, Double-blind, Multicenter, Placebo-controlled Phase III Clinical Study to Evaluate the Efficacy and Safety of SHR-1314 Injection in Adult Patients With Active Non-radiographic Axial Spondyloarthritis
Brief Title: A Trial of SHR-1314 Injection in Adult Patients With Active Non-radiographic Axial Spondyloarthritis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-1314-306
Record Dates: First submitted 2025-03-02; First posted 2025-03-06 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Active Non-radiographic Axial Spondyloarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-1314 Injection (Experimental): Subjects will receive SHR-1314 injection in the core treatment period and the extended treatment period.
  Interventions: Drug: SHR-1314 Injection
- SHR-1314 Placebo Injection (Placebo Comparator): Subjects will receive SHR-1314 placebo injection in the core treatment period and receive SHR-1314 injection in the extended treatment period.
  Interventions: Drug: SHR-1314 Injection; Drug: SHR-1314 Placebo Injection

INTERVENTIONS:
Drug: SHR-1314 Injection — SHR-1314 injection.
Drug: SHR-1314 Placebo Injection — SHR-1314 placebo injection.
  Arms: SHR-1314 Placebo Injection

SUMMARY:
The study is being conducted to evaluate the efficacy and safety of SHR-1314 injection in adult patients with active non-radiographic axial spondyloarthritis.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at the time of signing the informed consent form, regardless of gender.
2. BMI (Body Mass Index) ≥ 18 kg/m² at the time of screening.
3. Presence of objective signs of inflammation at the time of screening.
4. The subject voluntarily signs the ICF (informed consent form) before the start of any study-related procedures.
5. The subject is able to communicate effectively with the investigator, understands and is willing to strictly adhere to the requirements of the clinical study protocol to complete the study.

Exclusion Criteria:

1. Subjects with active systemic infection or severe infection.
2. Subjects with active tuberculosis or latent tuberculosis infection.
3. Subjects with lymphoma or lymphoproliferative disease.
4. Subjects with uncontrolled hypertension.
5. Subjects with history of malignancy within the past 5 years or current malignancy.
6. Subjects with moderate to severe congestive heart failure.
7. Subjects with history of organ transplantation, or severe, progressive, or uncontrolled diseases of any organ system.
8. Presence of protocol-defined abnormalities in laboratory tests and/or 12-lead ECG at the time of screening.
9. Pregnant or breastfeeding women.
10. known allergy to the study drug or any of its components.
11. Subjects with history of alcohol abuse or illegal drug use within the past year.
12. Receipt of a live vaccine within 12 weeks before randomization, or plans to receive a live vaccine during the study period.
13. Blood donation of approximately 500 mL within 8 weeks before randomization, or plans to donate blood during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants achieving ASAS 40 (ankylosing spondylitis disease activity score). | At the 16th week after administration.

SECONDARY OUTCOMES:
Proportion of participants achieving ASAS 20 (ankylosing spondylitis disease activity score). | At the 16th week after administration.
Change in CRP (C-reactive protein) value from baseline. | At the 16th week after administration.
AEs (adverse events). | Up to 60 weeks after administration.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided